| NCT04823624 |
|-------------|



Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS Version: 1.31.2020

**Protocol Title:** TIM3 Inhibition with MBG453 for Patients with Lower Risk MDS: an Adaptive Two-Stage Phase II Clinical Trial

#### **DF/HCC Principal Investigators/ Institutions:**

Andrew Brunner, MD/Massachusetts General Hospital Marlise Luskin, MD/Dana Farber Cancer Institute

#### **Main Consent**

#### INTRODUCTION AND KEY INFORMATION

All research is voluntary. It is your choice whether you take part in this research or not. If you decide to participate, please sign and date at the end of this form. We will give you a copy and you can refer to this consent form at any time.

The following is a short summary of this research study to help you decide whether you would like to be a part of this study. More detailed information is provided later in this form.

For purposes of this research, you will be referred to as a "participant."

#### 1. Why am I being invited to take part in a research study?

You are invited to take part in in this research study because you have lower risk myelodysplastic syndromes (MDS).

#### 2. Why is this research being done?

This research is being done to see how a study drug works in people with MDS.

#### 3. Who is supporting this research?

Novartis, a pharmaceutical company, is supporting this research study by providing funding for this study, including the study drug. The sponsor of the research is the DF/HCC.

#### 4. What does this research study involve and how long will it last?

The name of the study drug involved in this study is MBG453.


| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| 1/22/2024 | 12:08 PM |
|-----------|----------|

# NCT04823624


#### **Research Consent Form**

Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

The research study procedures include screening for eligibility and study treatment, including evaluations and follow up visits.

You will receive study treatment for as long as you and your doctor believe you are benefiting from the study drug. You will then be followed for 12 months after your last dose of the study drug or until you withdraw your consent to be contacted.

It is expected that about 20 people will take part in this research study.

Information about you and your health is personal and private. Generally, it cannot be obtained without your written permission. By signing this form, you are providing that permission and your information may be obtained and used in accordance with this informed consent and as required or allowed by law. This means that researchers may obtain information regarding your past medical history, as well as specimens and samples from previous health care providers such as hospitals and labs.

#### 5. What are the risks to participating in this study?

There are risks to taking part in any research study. We want to make sure you know about a few key risks right now. There may also be rare, serious and potentially life-threatening side effects. More detailed information is provided in the "What are the risks or discomforts of the research study?" section.

There is a risk that you could have side effects from the MBG453. These side effects may be worse and may be different than you would get with other approaches for your cancer.

Some of the most common side effects (happening in 10-30% of patients) that the study doctors know about are:

- Fatigue
- Headache
- Nausea
- Constipation
- Decreased appetite
- Shortness of breath
- Abdominal Pain
- Vomiting
- Diarrhea
- Joint aches


| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| 1/22/2024 12:08 PM | NCT04823624 |
|-----------------------|-------------|
| Pasaarch Consont Form | |

Dana-Farber/ Harvard Cancer Center

BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

 Low number of red blood cells, which may cause fatigue or shortness of breath

OHRS Version: 1.31,2020

- Low number of platelets, which may increase the risk of bleeding
- Low number of white blood cells, which may be a risk for infections such as pneumonia (infection of the lungs) or urinary tract infections.
- Fever, which may occur at the same time that the white blood cell count is low and require administration of antibiotics or admission to the hospital
- Swelling of the legs and ankles
- Dizziness

#### 6. Will being in this study benefit me in any way?

We do not know if taking part in this study will benefit you. This study may help researchers learn information that could help people in the future.

#### 7. What are my options?

Instead of being in this research study, you have other options which may include the following:

- Receive standard treatment including chemotherapies like azacitidine or decitabine, supportive transfusions, or growth factors
- Decide not to participate in this research study
- Participate in another research study.
- Receive no therapy specific to your cancer.
- Comfort care, also called palliative care. This type of care may help to reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly, but instead tries to treat the symptoms.

If you choose not to participate, are not eligible to participate, or withdraw from this research study, this will not affect your present or future care and will not cause any penalty or loss of benefits to which you are otherwise entitled.

We encourage you to take some time to think this over, to discuss it with other people and your primary doctor, and to ask questions at any time.

| Pag | $\sim$ | 2 | Λf | 21 |
|-----|--------|---|----|------------|
| гац | F | J | ΟI | <b>4</b> I |

| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| 1/22/2024 12:08 PM | NCT04823624 |
|-----------------------|-------------|
| Research Consent Form | |

#### A. WHY IS THIS RESEARCH STUDY BEING DONE?

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.


The U.S. Food and Drug Administration (FDA) has not approved MBG453 for your specific disease but it has been approved for other uses.

The study drug (MBG453) may interact with TIM-3 (an antibody which is a protein that attaches to foreign infectious/invading cells and signals the immune system) which might aid the immune system's (system in your body that fights against diseases) response by helping immune cells recognize, find, and destroy cancer cells in the body.

#### B. WHAT IS INVOLVED IN THE RESEARCH STUDY?

#### Before the research starts (screening):

After signing this consent form, you will be asked to undergo some screening tests or procedures to find out if you can be in the research study. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that you do not take part in the research study. If you have had some of these tests or procedures recently, they may or may not have to be repeated.

- A medical history, which includes questions about your demographics, health, current medications, and any allergies.
- **Physical Examination**, including the following:
  - Height/Weight/Body Surface Area Measurements. Height will only be measured at screening.
  - Blood Pressure
- Laboratory Tests, approximately <u>10</u> teaspoons/tablespoons of blood will be collected for the following purposes:
  - Routine clinical purposes, including a pregnancy test if you are a woman of childbearing potential.
  - Research testing.
- **Electrocardiogram (ECG)**, which measures your heart's electrical activity.
- **Measurement of vital signs**, which includes body temperature, pulse rate, and breathing rate.

| Page | 4 | of | 21 |
|------|---|----|----|

| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| /22/2024 12:08 PM | NCT04823624 |
|------------------------------------|-------------|
| Research Consent Form | |
| Dana-Farber/ Harvard Cancer Center | |

BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

• **Performance Status**, which evaluates how you are able to carry on with your usual activities.


If these tests show that you are eligible to participate in the research study, you may begin the study treatment. If you do not meet the eligibility criteria, you will not be able to participate in this research study.

## Additional research procedures to be performed at the time of screening but not required to determine eligibility:

 Bone marrow biopsy and/or aspirate, to evaluate the extent of your disease. For this test, a sample of bone marrow cells is taken by a needle inserted into a bone in your body. If a bone marrow biopsy is needed, a small piece of bone and the attached bone marrow is removed. These tests may be done under local anesthesia.

#### **Study Treatment Overview:**

Infused Study Drug: Each study treatment cycle last for 28 days (4 weeks) during this time you will be given MBG453 On Day 1 of each cycle into your vein (by intravenous infusion) over about 30 minutes. This will continue for as long as you are on the study.

#### Study Visit (Cycle 1 Day 1):

This visit will involve the following:

- MBG453 infusion.
- Medical History.
- Physical Exam.
- Laboratory Test, blood samples will be collected for routine clinical purposes.
- ECG
- Vital Signs Measurement.
- Performance Status.

#### Study Visit (Cycle 1 Days 8, 15, and 22):

This visit will involve the following:

- Medical History.
- Laboratory Test, blood samples will be collected for routine clinical purposes.
- Vital Signs Measurement.

#### Study Visit (Cycle 2 Day 1):


| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| 1/22/2024 12:08 PM | NCT04823624 |
|--------------------|-------------|

Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

#### This visit will involve the following:

- MBG453 infusion.
- Medical History.
- Physical Exam.
- Laboratory Test, blood samples will be collected for routine clinical purposes.


- Vital Signs Measurement.
- Performance Status.
- ECG

#### Study Visit (Cycle 2 Days 8, 15, and 22):

This visit will involve the following:

- Medical History.
- Laboratory Test, blood samples will be collected for routine clinical purposes.
- Vital Signs Measurement

#### Study Visit (Cycle 3 Day 1):

This visit will involve the following:

- MBG453 infusion.
- Medical History.
- Physical Exam.
- Laboratory Test, blood samples will be collected for routine clinical purposes.
- ECG
- Vital Signs Measurement.
- Performance Status.
- Bone Marrow Biopsy/Aspirate which will be used for analysis.

#### Study Visit (Cycle 3 Day 15):

This visit will involve the following:

- Medical History.
- Laboratory Test, blood samples will be collected for routine clinical purposes.
- Vital Signs Measurement.

#### **Study Visit (Cycle 4 Day 1):**

This visit will involve the following:

- MBG453 infusion.
- Medical History.


| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| 1/22/2024 12:08 PM | NCT04823624 |
|--------------------|-------------|

Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

- Physical Exam.
- Laboratory Test, blood samples will be collected for routine clinical purposes.


- ECG
- Vital Signs Measurement.
- Performance Status.

#### Study Visit (Cycle 4 Day 15):

This visit will involve the following:

- Medical History.
- Laboratory Test, blood samples will be collected for routine clinical purposes.
- Vital Signs Measurement

#### Study Visit (Cycles 5+ Day 1):

These visits will involve the following:

- MBG453 infusion.
- Medical History.
- Physical Exam.
- Laboratory Test, blood samples will be collected for routine clinical purposes.
- Vital Signs Measurement.
- Performance Status.
- ECG
- Bone Marrow Biopsy, which will be used for analysis.

#### Study Visit (End of Treatment):

This visit will occur 30 days after your last dose of the study drug and will involve the following:

- Medical History.
- Physical Exam.
- Laboratory Test, blood samples will be collected for routine clinical purposes.
- Vital Signs Measurement
- ECG
- Bone Marrow Biopsy, which will be used for analysis.

#### 

| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| 1 | 122 | /2024 | 12:08 | PМ |
|-----|-----|-------|-------|----|
| - 1 | 122 | 12024 | 12.00 | |

| NCT04823624 |
|-------------|

Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates


#### **Research Study Plan:**

| | Cycle 1 | | Cycle 2 | | | Cycles 3 | | Cycle 4 | | Cycle<br>5+ | End of<br>Treatment | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | Day<br>1 | Day<br>8 | Day<br>15 | Day<br>22 | Day<br>1 | Day<br>8 | Day<br>15 | Day<br>22 | Day 1 | Day<br>15 | Day<br>1 | Day<br>15 | Day<br>1 | 30 days<br>after last<br>dose |
| MBG453 | | Х | | | | Χ | | | | X | | Х | | х | |
| Medical<br>History | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х | Х |
| Physical<br>Exam | Х | Х | | | | X | | | | Х | | Х | | Х | Х |
| Laboratory<br>Test | Х | Χ | Х | Х | Х | X | X | X | Х | Χ | Х | X | Х | Х | Х |
| Vital Signs | Х | Χ | Х | Х | Х | Χ | Х | Х | X | X | X | Х | Х | X | X |
| Performance<br>Status | Х | Х | | | | Х | | | | Х | Х | | | | |
| ECG | Х | Х | | | | Χ | | | | Х | | Х | | Х | X |
| Bone Marrow<br>Biopsy/Aspir<br>ate | Х | | | | | | | | | Х | | | | х | Х |

#### **Planned Follow-up:**

We would like to keep track of your medical condition. Follow-up will be for 12 months from the last dose of the study drug. This will occur at approximately 30, 150, and 250 days after the last dose, and roughly 12 months from the last dose, and will be done in person or via phone/electronically. Keeping in touch with you and checking your condition helps us look at the long-term effects of the research study.

In addition, you can stop participating in the research study at any time, however, the FDA requires that any information collected up to the point of your withdrawal cannot be removed from the study.


| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| 1/22/2024 12:08 PM | NCT04823624 |
|----------------------------------------------------------|-------------|
| Research Consent Form Dana-Farber/ Harvard Cancer Center | |

#### C. WHAT ARE THE RISKS OR DISCOMFORTS OF THE RESEARCH STUDY?

BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

There are risks to taking part in any research study. One risk is that you may get a study drug that does not help treat your disease or that makes your condition or disease worse. Another risk is that there may be side effects.

All cancer treatments can have side effects, which can range from mild and reversible to severe, long lasting and possibly life-threatening. There is a great deal of variability among side effects of different cancer treatments and between individuals. In a research study, all of the risks or side effects may not be known before you start the study. You need to tell your doctor or a member of the study team immediately if you experience any side effects.

Everyone in the research study will be watched carefully for side effects. You will be monitored during the administration of study drugs to keep track of your blood counts and organ function, particularly your kidney and liver function. If you experience side effects, they may go away after you stop taking the study drug. Some side effects can be mild; but others can be long lasting and may never go away. Some may be life-threatening or fatal.

Since the effect of the study drug(s) taken with other medications may not be known, it is important that you tell the research doctor about all prescription and non-prescription drugs, herbal preparations and nutritional supplements that you are taking or planning to take. There may also be some foods that you should avoid while on this research study and your research doctor will review this information with you.

During the research study, you will be notified of newly discovered side effects or significant findings, which may affect your health or willingness to participate. You may be asked to sign a new consent form that shows that you have been informed of new information relating to this research study.

#### **Risks Associated with MBG453:**

#### Occasional (More than a 5% chance that this will happen):

- Constipation
- Abnormal physical weakness or lack of energy
- Fatigue
- Vomiting

#### Rare (Less than a 5% chance that this will happen):


| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| 1/22/2024 12:08 PM | NCT04823624 |
|--------------------|-------------|

Dana-Farber/ Harvard Cancer Center
BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

- Joint pain
- Cough
- Skin irritation (Dermatitis) possible symptoms include rash, itching, dry, cracked, or scaly skin, and swelling, burning or tenderness. This may require treatment with a topical medication or cream. Rarely it could require systemic treatment with a steroid.


- Dry skin
- Difficulty breathing
- Hypomagnesaemia or low levels of magnesium in the blood which could cause weakness and muscle cramping. Rarely heart rhythm abnormalities may occur. To treat this, you may need to get either oral or intravenous magnesium to replace these levels.
- Lethargy (fatigue/sleepiness)
- Chest pain
- Fluid in the lungs. Possible symptoms include wheezing or gasping for breath, difficulty breathing, and extreme shortness of breath that worsens with activity or when lying down. This can be dangerous if not evaluated and treated.
- Stomatitis or inflammation of the mucous membrane of the mouth which may be painful and cause difficulty swallowing.
- Abnormally rapid heart rate

#### Risks Associated with Bone Marrow Biopsies/Aspirations:

For this procedure, a numbing drug is injected into the skin over one of your hipbones. A needle is then inserted into the hipbones and a small piece of bone is removed (biopsy) or a sample of the bone marrow is removed (aspiration). The risks may include:

- Moderate pain and discomfort
- Bleeding at the biopsy/aspiration site
- Scarring at the biopsy/aspiration site
- Rarely, an infection at the biopsy/aspiration site
- Rarely, nerve injury at the biopsy/aspiration site

#### Reproductive Risks:

The drugs used in this research study may affect a fetus. While participating in this research study, and for at least 5 months after the last dose of the study drug, you should not:

- become pregnant
- nurse a baby
- father a baby


| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| 1/22/2024 12:08 PM | NCT04823624 |
|-----------------------|-------------|
| Research Consent Form | |

We can provide counseling about preventing pregnancy for either male or female study participants. Let your doctor know immediately if you become pregnant or find out that you are going to be the father of a child.

OHRS Version: 1.31,2020

If your partner becomes pregnant while you are on the study, it may be critical to share information regarding your participation in this research study with that person. Your research doctor should also be told if this happens.

#### Non-Physical Risks:

Because of side effects or the time required for tests and clinic visits while you are on this research study, you may be unable to keep up with your normal daily activities.

## D. WHAT WILL HAPPEN IF I AM REMOVED FROM THE STUDY OR DECIDE TO END MY PARTICIPATION IN THE RESEARCH?

You may be taken off the research study for any reason including:

- It is considered to be in your best interest
- The study treatment or procedures are found to be unsafe or ineffective
- There is any problem with following study treatments and procedures
- You are a female and become pregnant or plan to become pregnant
- Your condition worsens
- A decision is made to end the study
- Or for other unforeseen reasons that make it necessary to stop your participation in the research study

You can also choose to stop participating in the research study at any time. Tell the research doctor if you are thinking about stopping or decide to stop. He or she will tell you how to stop. Leaving the research study will not affect your medical care outside of the research study.

It is important to tell the research doctor if you are thinking about stopping so your research doctor can evaluate the risks from stopping the study drug.

It is important to note that although you may withdraw from study participation, the FDA requires that any information collected up to the point of your withdrawal cannot be removed from study records. Additionally, the research doctor may consult public records after you have withdrawn from the study.

#### 

| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| 1/22/2024 12:08 PM | NCT04823624 |
|----------------------------------------------------------|-------------|
| December Consent Form | |
| Research Consent Form Dana-Farber/ Harvard Cancer Center | |

#### E. WHAT ARE THE BENEFITS OF THIS RESEARCH STUDY?

BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

Taking part in this research study may or may not benefit you. We hope the information learned from this research study will provide more information about MBG453 and its effects on your disease.


#### F. WILL I BE PAID TO TAKE PART IN THIS RESEARCH STUDY?

You will not be paid for participating in this study.

We may use your samples and information to develop a new product or medical test to be sold. The sponsor and hospital may benefit if this happens. There are no plans to pay you if your samples are used for this purpose.

#### G. WHAT ARE YOUR COSTS?

Taking part in this research study may lead to added costs to you or your insurance company. This may mean that you need to make more visits to the

clinic or hospital than if you were getting the usual approach to treat your disease. You may:

- Have more travel costs
- Need to take more time off work
- Have other additional personal costs

You will not be charged for MBG453.

You or your insurance company will be charged for portions of your care during this research study that are considered standard care. Standard of care is the care that you would receive regardless of whether you were enrolled in the study or not. You may be responsible for co-payments, co-insurance, premiums and deductibles that are typical for your insurance coverage. This includes the cost of tests, procedures, or medicines to manage any side effects, unless you are told that certain tests, done for research only, are supplied at no charge.

If you have questions about your insurance coverage, or the items you might be required to pay for, please call financial services for information. The contact information for financial services are:

- Brigham and Women's Hospital: (617) 732-5524 or (617) 732-7485
- Dana-Farber Cancer Institute: (617) 632-3455


| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| 1/22/2024 12:08 PM | NCT04823624 | ] |
|---|---|---|
| Research Consent Form | | ] |
| Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners N | letwork Affiliates | OHRS Version: 1.31.2020 |

Massachusetts General Hospital: (617) 726-2191

The National Cancer Institute provides an online resource to help people participating in cancer clinical trials understand which services their insurance company is required by law to pay. This can be found at the website below or can be provided by the study team:

> www.cancer.gov or 1-800-4-CANCER (1-800-422-6237)

### H. WHAT HAPPENS IF I AM INJURED OR BECOME SICK BECAUSE I TOOK PART IN THIS RESEARCH STUDY?

If you think you have been injured as a result of taking part in this research study, tell the person in charge of this research study as soon as possible. The research doctor's name and phone number are listed in this consent form.

The treating hospital will offer you the care needed to treat injuries directly resulting from taking part in this research. These treatments may be billed to you or your insurance company. You will be responsible for deductibles, co-

payments and co-insurance. There are no plans to pay you or give you other compensation for the injury.

You do not give up your legal rights by signing this form.

We will need to collect certain personal information about you for insurance or payment reporting purposes, such as your name, date of birth, gender, social security number or Medicare identification number and information related to this research study. We may be required to report this information to the Centers for Medicare & Medicaid Services. We will not use this information for any other purpose.

If you go to the Emergency Room or to another hospital or doctor it is important that you tell them that you are in this research. If possible, you should give them a copy of this consent form.

#### 

| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| 1/22/2024 12:08 PM | NCT04823624 |
|------------------------------------|-------------|
| Research Consent Form | |
| Dana-Farher/ Harvard Cancer Center | |

BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

#### I. WHOM DO I CONTACT IF I HAVE QUESTIONS ABOUT THE RESEARCH STUDY?

If you have questions about the study, please contact the research doctor or study staff as listed below:

#### **Massachusetts General Hospital**

• Andrew Brunner, MD: 617-643-8690

#### **Dana-Farber Cancer Institute**

• Marlise Luskin, MD: 617-632-1906

24-hour contact: Please contact your hospital and ask that your doctor be paged:

- Massachusetts General Hospital at 617-724-4000
- Dana-Farber Cancer Institute: (617) 632-3455

For questions about your rights as a research participant, please contact a representative of the Office for Human Research Studies at Dana-Farber Cancer Institute (617) 632-3029. This can include questions about your participation in the study, concerns about the study, a research related injury, or if you feel/felt under pressure to enroll in this research study or to continue to participate in this research study.

#### J. RETURN OF RESEARCH RESULTS

Tests done on samples in this research study are only for research and have no clear meaning for your health care. For this reason, your study doctor will not share the results with you.

#### K. CLINICALTRIALS.GOV (CT.GOV)

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This web site will not include information that can identify you. At most, the web site will include a summary of the results. You can search this web site at any time.

#### L. FUTURE USE OF DATA AND SPECIMENS

Your personal information and/or biospecimens collected during this study may be stored and used for future research. Any personal identifiers will be removed, 

| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |



| NCT04823624 |
|-------------|

#### **Research Consent Form**

Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

before they are shared, so that the information or samples cannot be linked back to you.

Investigators, including investigators from collaborating institutions, can request this data and samples for new research. Samples and data may also be shared with outside non-profit academic investigators as well as with for-profit pharmaceutical investigators or commercial entities, with whom we collaborate.

You will not be asked to provide additional informed consent for the use of your identifiable information or samples in future research.

Future research studies may include genetic research. Your genes are unique to you. At this time, you cannot be identified through this research, if the samples and specimens are de-identified. There is a risk that you might be reidentified in the future as genetic research progresses

#### M. CONFIDENTIALITY

We will take measures to protect the privacy and security of all your personal information, but we cannot guarantee complete confidentiality of study data.

Medical information created by this research study may become part of your hospital medical record and may be forwarded to your primary doctor. Information that does not become part of your medical record will be stored in your study file. It may also become part of a research database.

Participation in this study involves providing a specimen of your tissue; please know that if the research doctor leaves the institution, the research and the tissue might remain at the research doctor's current institute or might be transferred to another institution.

The study team plans to publish the results of this research study and when we do, we may be asked to make the data we collect available to other researchers. We will not include information that identifies you in any publications or to the researchers who request the data to do additional research.

Your de-identified specimens or genetic data may also be placed into one or more publicly-accessible scientific databases. Through such databases, researchers from around the world will have access to de-identified samples or data for future research.

#### 

| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| 1/22/2024 12:08 PM | NCT04823624 |
|-----------------------|-------------|
| Research Consent Form | |

There is a risk that deidentified research data that is shared with outside collaborators may be reidentified. When deidentified data and specimens are shared with outside collaborators agreements limit what the outside collaborators can do with the information to help prevent reidentification.


#### N. FINANCIAL DISCLOSURES

It is possible that certain researchers on this study may have earned money from, or own some publicly-traded stock in, the company that makes or is developing the study drug. The amount of money that a researcher may earn and still take part in research is limited by the Harvard Medical School Faculty of Medicine Policy on Conflicts of Interest and Commitment. If you have further questions, please speak with a member of the study team or contact the Dana-Farber Cancer Institute Office of Research Integrity at 617-432-4557 or researchintegrity@dfci.harvard.edu.

Dana-Farber Cancer Institute has a financial interest in the investigational compound used in this trial, MBG453. This financial interest could be affected by the outcome of this research. Additional information is provided in the Patient Information Sheet available to participants.

#### O. GENETIC RESEARCH

This research will involve genomic testing.

The Genetic Information Nondiscrimination Act of 2008 (GINA) is a federal law that protects Americans from being treated unfairly because of differences in their DNA that may affect their health, and may prevent discrimination by health insurers and employers based on genetic information. GINA is intended to ease concerns about discrimination that might keep some people from getting genetic

tests that could benefit their health, and enable people to take part in research studies such as this without fear that their DNA information might be used against them by health insurers or their workplace. This protection does not extend to disability or life insurance. Additional information can be found at <a href="http://www.genome.gov/10002328">http://www.genome.gov/10002328</a>.

#### P. PRIVACY OF PROTECTED HEALTH INFORMATION (HIPAA AUTHORIZATION)

The Health Insurance Portability and Accountability Act (HIPAA) is a federal law that requires Dana-Farber/Harvard Cancer Center (DF/HCC) and its affiliated research doctors, health care providers, and physician network to protect the


| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| 1/22/2024 12:08 PM | NCT04823624 |
|-----------------------|-------------|
| Research Consent Form | |

privacy of information that identifies you and relates to your past, present, and future physical and mental health conditions ("protected health information"). If you enroll in this research study, your "protected health information" will be used and shared with others as explained below.


### 1. What protected health information about me will be used or shared with others during this research?

- Existing medical records, including mental health records.
- New health information created from study-related tests, procedures, visits, and/or questionnaires

#### 2. Why will protected information about me be used or shared with others?

The main reasons include the following:

- To conduct and oversee the research described earlier in this form;
- To ensure the research meets legal, institutional, and accreditation requirements;
- To conduct public health activities (including reporting of adverse events or situations where you or others may be at risk of harm); and
- To provide the study sponsor with information arising from an adverse event or other event that relates to the safety or toxicity of the drug(s) used in the study and for the purpose of this or other research relating the study drug(s) and their use in cancer;
- To better understand the diseases being studied and to improve the design of future studies; and,
- Other reasons may include for treatment, payment, or health care operations. For example, some medical information produced by this research study may become part of your hospital medical record because the information may be necessary for your medical care. (You will also be given a notice for use and sharing of protected health information.)

#### 3. Who will use or share protected health information about me?

 DF/HCC and its affiliated research doctors and entities participating in the research will use and share your protected health information. In addition, other DF/HCC offices that deal with research oversight, billing or quality assurance will be able to use and share your protected health information.

| Page ' | 17 c | of 21 |
|--------|------|-------|
|--------|------|-------|

| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| 1/22/2024 12:08 PM | NCT04823624 |
|-----------------------|-------------|
| Research Consent Form | |

### 4. With whom outside of DF/HCC may my protected health information be shared?

While all reasonable efforts will be made to protect the confidentiality of your protected health information, it may also be shared with the following entities:


- Outside individuals or entities that have a need to access this information to perform functions relating to the conduct of this research such as analysis by outside laboratories on behalf of DF/HCC and its affiliates (for example, data storage companies, insurers, or legal advisors).
- The sponsor(s) of the study, its subcontractors, representatives, business partners, and its agent(s): DF/HCC
- Other research doctors and medical centers participating in this research, if applicable
- Federal and state agencies (for example, the Department of Health and Human Services, the Food and Drug Administration, the National Institutes of Health, and/or the Office for Human Research Protections), or other domestic or foreign government bodies if required by law and/or necessary for oversight purposes. A qualified representative of the FDA and the National Cancer Institute may review your medical records.
- Hospital accrediting agencies
- A data safety monitoring board organized to oversee this research, if applicable
- Other, the funder(s) of the study, its subcontractors, representatives, business partners, and its agent(s): Novartis

Some who may receive your protected health information may not have to satisfy the privacy rules and requirements. They, in fact, may share your information with others without your permission.

### 5. For how long will protected health information about me be used or shared with others?

 There is no scheduled date at which your protected health information that is being used or shared for this research will be destroyed, because research is an ongoing process.

#### 6. Statement of privacy rights:

 You have the right to withdraw your permission for the research doctors and participating DF/HCC entities to use or share your protected health information. We will not be able to withdraw all the information that 

| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| 1/22/2024 12:08 PM | NCT04823624 | _ |
|--------------------------|-------------|---|
| December October 5 Forms | | |

Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

already has been used or shared with others to carry out related activities such as oversight, or that is needed to ensure quality of the study. To withdraw your permission, you must do so in writing by contacting the researcher listed above in the section: "Whom do I contact if I have questions about the research study?"


 You have the right to request access to your protected health information that is used or shared during this research and that is related to your treatment or payment for your treatment, but you may access this information only after the study is completed. To request this information, please contact the researcher listed above in the section: "Whom do I contact if I have guestions about the research study?"

| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| I/22/2024 12:08 PM | NCT04823624 | |
|---|---|---|
| Research Consent Form Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners N | Network Affiliates | OHRS Version: 1.31.2020 |
| Q. DOCUMENTATION OF CONSENT | | |
| <ul><li>participating in this study</li><li>I have had all of my que</li><li>I am willing to participate</li></ul> | stions answered to my sati | isfaction; |
| Signature of Participant or Legally Authorized Representat | Date tive | |

Relationship of Legally Authorized Representative to Participant


| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |

| 1/22/2024 | 12:08 PM |
|-----------|----------|
|-----------|----------|

| NCT04823624 |
|-------------|

### **Research Consent Form**

Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

| | To be completed by person obtaining consent: |
|---|---|
| | Adult Participant |
| The c | onsent discussion was initiated on (date). |
| Signa | ture of individual obtaining consent: |
| Printe | d name of above: |
| Date: | |
| | copy of this signed consent form will be given to the participant or legally authorized epresentative. |
| □ 1) | The participant is an adult and provided consent to participate. |
| | 1a) Participant (or legally authorized representative) is a non-English speaker and signed the translated Short Form in lieu of English consent document: |
| in | As someone who understands both English and the language used by the participant, I terpreted and/or witnessed, in the participant's language, the researcher's presentation of e English consent form. The participant was given the opportunity to ask questions. |
| | Signature of Interpreter/Witness: |
| | Printed Name of Interpreter/Witness: |
| | Date: |
| | 1b) Participant is physically unable to sign the consent form because: |
| | ☐ The participant is illiterate. |
| | ☐ The participant has a physical disability. |
| | Other (please describe): |
| | The consent form was presented to the participant who was given the opportunity to ask questions and who communicated agreement to participate in the research. |
| | Signature of Witness: |
| | Printed Name of Witness: |
| | Date: |
| | The participant is an adult who lacks capacity to provide consent and his/her legally uthorized representative: |
| | 2a) gave permission for the adult participant to participate |
| ☐ 2h | b) did not give permission for the adult participant to participate |


| DFCI Protocol Number: 20-637 | Approved Date (DFCI IRB Approval): 10/04/2022 |
|---|---|
| Date Posted for Use: 10/05/2022 | |